CLINICAL TRIAL: NCT06670612
Title: The Effect of Nature-Based Music Concert on Pain and Physiological Parameters in Intensive Care Patients
Brief Title: The Effect of Nature-Based Music Concert on Intensive Care Patients
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sevcan Karataş (Other)
Responsible Party: Sponsor-Investigator, Sevcan Karataş, assistant professor, İstanbul Yeni Yüzyıl Üniversitesi
Organization: İstanbul Yeni Yüzyıl Üniversitesi (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 2024/03-1241
Record Dates: First submitted 2024-10-30; First posted 2024-11-01 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Patient Care; Patient Care in ICU
Keywords: music; pain; nature based music; physiological parameter
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): . Being 18 years or older
  * Having orientation to place and time
  * No communication (visual, auditory) barriers
  * No neuromuscular blockade with medication
  * Not applying nerve block,
  * Not having peripheral neuropathy or quadriplegia
  * Sedation level 1, 2, 3 and 4 according to the Ramsey Sedation Scale (RSS)
  Interventions: Other: nature based music concert
- control group (No Intervention): . Being 18 years or older
  * Having orientation to place and time
  * No communication (visual, auditory) barriers
  * No neuromuscular blockade with medication
  * Not applying nerve block,
  * Not having peripheral neuropathy or quadriplegia
  * Sedation level 1, 2, 3 and 4 according to the Ramsey Sedation Scale (RSS)

INTERVENTIONS:
Other: nature based music concert — It will be a resource for healthcare professionals to develop a behavior that will support patients in intensive care in relieving their pain and stabilizing their physiological parameters with nature-based music, and will contribute to the literature.
  Other Names: music concert
  Arms: intervention group

SUMMARY:
Purpose: This study was planned to determine the effect of nature-based music recital on pain and physiological parameters in intensive care patients.

Design: This research will be conducted as a pre-test post-test randomized controlled intervention study. Patient Information Form, Numerical Pain Scale and Physiological Parameters Tracking Form will be used as data collection forms.

H1: Nature-based music recital has an effect on pain level

H2: Nature-based music recital has an effect on physiological parameters

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years or older
* Having orientation to place and time
* No communication (visual, auditory) barriers
* No neuromuscular blockade with medication
* Not applying nerve block,
* Not having peripheral neuropathy or quadriplegia
* Sedation level 1, 2, 3 and 4 according to the Ramsey Sedation Scale (RSS)

Exclusion Criteria:

* Glasgow Coma Scale score below 13 points
* Being diagnosed with a psychiatric disease
* Having dementia/brain dysfunction
* Having a hearing-related anomaly or health problem
* The patient has not undergone any painful procedure within the last hour.
* Sedation level should be 5 and 6 according to RSQ

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2024-04-10 (Actual); Primary Completion 2024-11-10 (Estimated); Study Completion 2025-04-10 (Estimated)

PRIMARY OUTCOMES:
Numerical Pain Scale | 1 hour from the music concert to the end of the application
  The numerical scale, which is the most commonly used scale in diagnosing pain, is quite simple to use. This scale has numerical values between 0 and 10 points, and the individual is shown the scale and asked to choose the number that best describes the pain. It consists of a horizontal line with a starting point of "0" or "No pain" and an end point of "10" or "Unbearable pain".
Physiological Parameters Tracking Form | 1 hour from the music concert to the end of the application
  It is a form containing patients' physiological parameters. While the patients are lying down in their rooms, blood pressure will be measured from the brachial artery, and heart rate and oxygen saturation values will be measured by the researcher using bedside monitors with pulse oximeter sensors.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Yeni Yuzyil University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No